CLINICAL TRIAL: NCT06316258
Title: Evaluating the Feasibility and Acceptability of Compassion Focused Therapy Group Intervention for Adults With Moderate-severe Acquired Brain Injury in an Inpatient Neurorehabilitation Setting
Brief Title: Evaluating a CFT Group for Adults With Acquired Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 333112
Record Dates: First submitted 2024-02-01; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Acquired Brain Injury Including Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassion focused therapy group (Experimental): 6 week compassion focused therapy group for adults with ABI
  Interventions: Behavioral: Compassion focused therapy group

INTERVENTIONS:
Behavioral: Compassion focused therapy group — 6 session compassion focused therapy group for adults with ABI

SUMMARY:
Emotional difficulties such as anxiety and depression are common after experiencing a brain injury. The compassion focused therapy (or CFT) model proposes the importance of developing skills in being able to self-soothe and be self-compassionate to counteract feelings of distress. Several studies have shown that therapy groups using CFT techniques are helpful, but there has only been one previous study of a CFT group with people with acquired brain injury. This study aims to evaluate a new CFT group for people who have had a brain injury and are currently receiving inpatient neuro-rehabilitation. The group will have six weekly sessions with 4-6 people in each group. The group will be run at the inpatient neuro-rehabilitation unit. As this is a new group that has not been run before, it will be a small study to see whether the group is feasible and acceptable to attendees. The study will evaluate whether the group can be run as planned and how many people attend. The investigators will also interview people who attended the group to find out what they thought of the group.

The study also aims to use four questionnaires measuring emotional distress, well-being, self-compassion and quality of life to measure the effect of the group. Group attendees questionnaire scores from before and after the group will be compared to see if there has been any change due to attending the group.

This project is being completed as part of a Doctorate in Clinical Psychology at King's College London, and will be recruiting patients from an inpatient neurorehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

1. Has experienced a non-progressive acquired brain injury
2. Is at least 18 years old
3. Has capacity to consent to take part in the group and associated research project
4. Is currently experiencing emotional distress, as identified descriptively by the treating team and indicated by a minimum score of 8 or above (mild symptoms) on the HADS.

Exclusion Criteria:

1. Has a [severe] cognitive impairment to a degree that this is considered by the treating team to prevent their ability to participate in the group despite adaptations.
2. Has a [severe] communication impairment to a degree that is considered by the treating team to prevent their ability to participate in or understand the group content despite adaptations.
3. Is currently experiencing a severe mental health disorder or crisis that would impact on their ability to participate in the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Demand - patients referred and screened for the group | At screening/enrollment
  Number of patients referred and screened
Demand - patients recruited | At screening/enrollment
  Number of patients recruited to group
Demand - attendance | Weeks 1-6 at each weekly group session
  Session attendance rate
Implementation - patients per group | Weeks 1-6 at each weekly group session
  Number of patients per group
Implementation - group sessions completed | Weeks 1-6 at each weekly group session
  Number of group sessions completed out of 6
Implementation - practice sessions completed | Weeks 1-6 at each weekly group session
  Number of additional practice sessions completed out of 6
Practicality - delivery of intervention | Weeks 1-6 at each weekly group session
  The number of items covered in the session out of the items that were planned in the session guide
Acceptability - end of session ratings scores | Weeks 1-6 at each weekly group session
  Patient ratings of enjoyment, understanding and helpfulness using 'Session Rating Form' designed for study
Acceptability - patient interview feedback | Interview time point after week 6
  Feedback from attendees collected via recorded semi-structured interviews after end of intervention

SECONDARY OUTCOMES:
Change in emotional distress questionnaire score | 2-week Baseline, week 1 (pre-group), week 6 (post-group), 2-week follow-up
  Measured using Hospital Anxiety Depression Scale (HADS)
Change in mental well-being questionnaire score | 2-week Baseline, week 1 (pre-group), week 6 (post-group), 2-week follow-up
  Measured using Warwick Edinburgh Mental Well-Being Scale (WEMWBS)
Change in self-compassion questionnaire score | 2-week Baseline, week 1 (pre-group), week 6 (post-group), 2-week follow-up
  Measured using Self-Compassion Scale Short Form (SCS-SF)
Change in quality of life questionnaire score | 2-week Baseline, week 1 (pre-group), week 6 (post-group), 2-week follow-up
  Measured using Quality of Life after Brain Injury Overall Scale (QOLIBRI-OS)